CLINICAL TRIAL: NCT05030142
Title: Evaluation of Mechanical Thrombectomy in Acute Ischemic Stroke Related to a Distal Arterial Occlusion: a Randomized Controlled Trial
Brief Title: Evaluation of Mechanical Thrombectomy in Acute Ischemic Stroke Related to a Distal Arterial Occlusion
Acronym: DISCOUNT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: APHP200028; 2021-A00516-35 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-07-31; First posted 2021-09-01 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acute Ischemic Stroke (AIS) Related to a Distal Occlusion
Keywords: Acute Ischemic Stroke; Distal occlusions; Mechanical Thrombectomy
MeSH Terms: conditions — Ischemic Stroke | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanical thrombectomy (Experimental): Mechanical thrombectomy (using a stent retriever among the following:Trevo NXT ProVue Retriever, Catchview mini, pReset Lite, Tigertriever 13) in association with the best medical treatment (usual care)
  Interventions: Procedure: Mechanical Thrombectomy
- Active Comparator (Active Comparator): Best medical treatment alone (usual care)
  Interventions: Drug: Best medical treatment alone

INTERVENTIONS:
Procedure: Mechanical Thrombectomy — Mechanical thrombectomy (using a stent retriever among the following:Trevo NXT ProVue Retriever, Catchview mini, pReset Lite, Tigertriever 13) in association with the best medical treatment (usual care)
  Other Names: Experimental group
  Arms: Mechanical thrombectomy
Drug: Best medical treatment alone — Best medical treatment alone (usual care)
  Other Names: Control group
  Arms: Active Comparator

SUMMARY:
Mechanical thrombectomy (MT) has shown its effectiveness for the treatment of acute ischemic stroke (AIS) related to large vessel occlusion and rapidly became a cornerstone in the management of these patients. No strong evidence is available on the benefit of MT in AIS related to more distal occlusions. Some previous observational studies suggested a possible benefit but most of them were single-centre and retrospective studies providing a very low level of evidence. To date, no randomized controlled trial has been conducted in this indication, which represents 10% to 20% of all AIS involving intracranial vessel occlusions.

This research is a multicenter open randomized controlled trial with two parallel groups : best medical treatment alone VS mechanical trombectomy + best medical treatment.

DETAILED DESCRIPTION:
The main objective of this trial is to assess the efficacy of mechanical thrombectomy in addition to the best medical treatment as compared to the best medical treatment alone in AIS related to a distal intracranial artery occlusion. The medical device used will be a stent retriever among : Trevor NXT ProVue Retriever ; Catchview mini ; pReset Lite ; Tigertriever13, and the medical treatment used will depend on the stroke's etiology and will consist of IV trhombolysis or tenecteplase or antiplatelet therapy or anticoagulant therapy ... The main inclusion criteria are : 1) patients aged ≥ 18 years ; 2) Delay between symptoms onset and expected groin puncture ≤ 6h ; 3) Symptomatic occlusion as evaluated by a National Institute of Health Stroke Score (NIHSS) ≥ 5 ; 4) Distal occlusion evaluated on CT angiography (CTA) or magnetic resonance imaging (MRI) and defined as an occlusion in one of the following segments : a-Distal M2, above the mid-height of the insula, b-M3 segment, c-Posterior cerebral artery (PCA) = P1, P2 or P3 segment, d-Anterior cerebral artery (ACA) : A1, A2 or A3 segment ; 5) Written informed consent signed by the patient or the trustworthy person / family member / close relative, or inclusion in case of emergency and written informed consent will be signed by the patient (if needed by trustworthy person, family member or close relative) as soon as possible (article L1122-1-2 of the French Public Health Code).

The secondary objectives and endpoints are to evaluate the : 1) Success of the procedure defined as recanalization of the occluded vessel, evaluated on the AOL (Arterial Occlusion Lesion) score within 48 hours ; 2) Excellent clinical outcome (defined as a modified Rankin scale [mRS]≤1) at 3 months ; 3) Safety with reporting of all adverse and serious adverse events with a particular attention to perforation rate, embolus migration in a new territory and symptomatic hemorrhagic complications ; 4) Death rate up to 3 months ; 5) Cost effectiveness and utility of the procedure. The study will also evaluate the rate of angiographic reperfusion in the intervention group on the final angiogram at the end of the MT (which is part of the intervention) using the modified thrombolysis in cerebral infarction (mTICI) (2B-3) and the eTICI.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Delay between symptoms onset and expected groin puncture ≤ 6 h
* Symptomatic occlusion as evaluated by a National Institute of Health Stroke Score (NIHSS) ≥ 5
* Distal occlusion evaluated on CT angiography (CTA) or magnetic resonance imaging (MRI) and defined as an occlusion in one of the following segments:

  * Distal M2, above the mid-height of the insula
  * M3 segment
  * Posterior cerebral artery (PCA): P1, P2, P3 segments
  * Anterior cerebral artery (ACA): A1, A2, A3 segments
* Written informed consent signed by the patient or the trustworthy person / family member / close relative, or inclusion in case of emergency and written informed consent will be signed by the patient (if needed by trustworthy person, family member or close relative) as soon as possible (article L1122-1-2 of the French Public Health Code)

Exclusion Criteria:

* Pregnancy or breastfeeding woman
* Contra-indication for femoral, radial or humeral arterial puncture
* Tandem occlusion (i.e.: concomitant cervical and intra-cranial arterial occlusion)
* Allergy to iodinated contrast media
* Known renal insufficiency (confirmed by previous result of creatinine clearance < 30 ml/min)
* Secondary distal occlusion (i.e., complicating a MT for a proximal occlusion, or any other endovascular intracranial procedure)
* Aortic dissection
* Asymptomatic or minor stroke (i.e.: NIHSS < 5)
* Pretreatment mRS > 1 (pre-stroke)
* Anticipated limitations for anesthesia
* Participation in another trial (Jardé 1 and Jardé 2)
* Absence of affiliation to National French social security system
* Under legal protection measure (tutorship or curatorship) and patient deprived of freedom
* A pre-existing hemorrhage in the brain tissue fed by the target vessel
* Known hypersensitivity to nickel/titanium
* Stenosis and/or with a stent proximal to the site of the thrombus which could preclude the retrieval of the stent retriever
* Angiographic evidence of carotid dissection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Estimated)
Dates: Start 2021-11-14 (Actual); Primary Completion 2024-02-14 (Estimated); Study Completion 2024-02-14 (Estimated)

PRIMARY OUTCOMES:
Good clinical outcome (defined as a modified Rankin Scale [mRS] ≤ 2) | At 3 months
  mRS of 0-2 (evaluated by an independent assessor blinded to the intervention received by the patient)

SECONDARY OUTCOMES:
Recanalization of the occluded vessel | 48 hours after the mechanical thrombectomy
  Evaluation of AOL (Arterial Occlusion Lesion scale) ≥ 2 on vascular brain imaging (magnetic resonance MR) or computed tomography (CT) angiography in patients belonging to both arms
Angiographic reperfusion in the intervention group | End of the mechanical thrombectomy procedure
  Use of the mTICI score (successful reperfusion: mTICI 2b-3) and the eTICI (extended thrombolysis in cerebral infarction) score (successful reperfusion: eTICI ≥ 2b67) on the control digital subtraction angiography (DSA)
Excellent Clinical outcome (defined as a modified Rankin Scale [mRS] ≤ 1) | At 3 months
  mRS of 0-1 (evaluated by an independent assessor blinded to the intervention received by the patient)
Perforation rate | End of mechanical thrombectomy procedure
  Defined as contrast material extravasation either on digital subtraction angiography [DSA] or control CT scan
Embolus migration in a new territory | End of mechanical thrombectomy procedure
  evaluated on digital subtraction angiography [DSA]
Symptomatic intracranial hemorrhage | within 7 days
  evaluated on CT-scan or MRI according to the ECASS II criteria
Subarachnoid hemorrhage | within 48 hours
  evaluated on CT-scan or MRI and define as the abnormal presence of blood within the subarachnoid space presence of blood within the subarachnoid space
Safety : incidence of adverse events | At 3 months
  Reporting of all adverse events
Safety : incidence of serious adverse events | At 3 months
  Reporting of all serious adverse events
Death rate | At 3 months
  Mortality
Utility of the procedure | At 3 months
  Incremental cost utility ratio
Cost effectiveness | At 3 months
  Cost per additional survivor (health-economics analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric Clarençon, Professor, Principal Investigator — APHP
Locations (1):
- Frédéric CLARENCON, Paris, France

IPD SHARING:
Plan to Share IPD: Yes
Data are available upon reasonable request. The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients. Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal.

REFERENCES:
- [Derived] Clarencon F, Durand-Zaleski I, Premat K, Baptiste A, Chabert E, Ferrier A, Labeyrie MA, Reiner P, Spelle L, Denier C, Tuilier T, Hosseini H, Rodriguez-Regent C, Turc G, Fauche C, Lamy M, Lapergue B, Consoli A, Barbier C, Boulanger M, Bricout N, Henon H, Gory B, Richard S, Rouchaud A, Macian-Montoro F, Eker O, Cho TH, Soize S, Moulin S, Gentric JC, Timsit S, Darcourt J, Albucher JF, Janot K, Annan M, Pico F, Costalat V, Arquizan C, Marnat G, Sibon I, Pop R, Wolff V, Shotar E, Lenck S, Sourour NA, Radenne A, Alamowitch S, Dechartres A. Evaluation of mechanical thrombectomy in acute ischemic stroke related to a distal arterial occlusion: A randomized controlled trial. Int J Stroke. 2024 Mar;19(3):367-372. doi: 10.1177/17474930231205213. Epub 2023 Oct 12. PMID 37740419